CLINICAL TRIAL: NCT01777282
Title: A 52-Week, Open-Label, Multicenter Study to Determine the Long Term Safety and Efficacy of Albiglutide in Combination With Monotherapy of Oral Antihyperglycemic Medications in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Determine the Long Term Safety and Efficacy of Albiglutide in Combination With Oral Monotherapy Antihyperglycemic Medications in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116170
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus
Keywords: albiglutide; Japanese; glucagon-like peptide-1; GSK716155
MeSH Terms: conditions — Diabetes Mellitus | interventions — rGLP-1 protein; Sulfonylurea Compounds; Biguanides; 2,4-thiazolidinedione; Glycoside Hydrolase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Albiglutide + Sulfonylurea (Active Comparator): Albiglutide in combination with background sulfonylurea
  Interventions: Drug: Albiglutide; Drug: Sulfonylurea
- Albiglutide + Biguanide (Active Comparator): Albiglutide in combination with background biguanide
  Interventions: Drug: Albiglutide; Drug: Biguanide
- Albiglutide + Glinide (Active Comparator): Albiglutide in combination with background glinide
  Interventions: Drug: Albiglutide; Drug: Glinide
- Albiglutide + Thiazolidinedione (Active Comparator): Albiglutide in combination with background thiazolidinedione
  Interventions: Drug: Albiglutide; Drug: Thiazolidinedione
- Albiglutide + Alpha-glucosidase inhibitor (Active Comparator): Albiglutide in combination with background alpha-glucosidase inhibitor
  Interventions: Drug: Albiglutide; Drug: Alpha-glucosidase inhibitor

INTERVENTIONS:
Drug: Albiglutide — Albiglutide is a fixed-dose, fully disposable pen injector system for delivery of albiglutide from a prefilled dual chamber glass cartridge that is an integral part of the pen. It is intended for single use by the subject. It is designed for manual reconstitution of the dose, priming, and insertion of the pen needle, and manual injection by the subject. The subject will inject albiglutide 30 mg weekly for 52 weeks (with optional uptitration to 50 mg weekly) subcutaneously into the abdomen, alternating between left and right sides. The pen is designed to work with standard pen needles.
Drug: Sulfonylurea — Single oral antidiabetic drug as a background therapy, to be continued as previously prescribed.
  Arms: Albiglutide + Sulfonylurea
Drug: Biguanide — Single oral antidiabetic drug as a background therapy, to be continued as previously prescribed.
  Arms: Albiglutide + Biguanide
Drug: Glinide — Single oral antidiabetic drug as a background therapy, to be continued as previously prescribed.
  Arms: Albiglutide + Glinide
Drug: Thiazolidinedione — Single oral antidiabetic drug as a background therapy, to be continued as previously prescribed.
  Arms: Albiglutide + Thiazolidinedione
Drug: Alpha-glucosidase inhibitor — Single oral antidiabetic drug as a background therapy, to be continued as previously prescribed.
  Arms: Albiglutide + Alpha-glucosidase inhibitor

SUMMARY:
This study is designed to examine the long term safety and efficacy of weekly subcutaneously injected albiglutide in combination with a single oral antidiabetic drug for 52 weeks in Japanese subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This study is designed to examine the long term safety and efficacy of weekly subcutaneously injected albiglutide in combination with a single oral antidiabetic drug for 52 weeks in Japanese subjects with type 2 diabetes mellitus. Subjects with a historical diagnosis of type 2 diabetes mellitus who are inadequately controlled on a single oral antidiabetic agent will be recruited into the study. Subjects will continue on their single antidiabetic agent and once weekly albiglutide will be added.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of Type 2 Diabetes Mellitus, who are experiencing inadequate glycemic control and receiving treatment with a stable dose of a single oral antidiabetic medication
* Body mass index (BMI) 17 to 40 kg/ m2 inclusive
* Subjects with an HbA1c between 7.0% and 10.0% at Screening
* Creatinine clearance >30 mL/min (calculated using the Cockcroft-Gault formula)

Exclusion Criteria:

* History of type 1 diabetes mellitus
* Female subject is pregnant, lactating, or <6 weeks postpartum
* Clinically significant cardiovascular and/or cerebrovascular disease
* Current ongoing symptomatic biliary disease, clinical signs or symptoms of pancreatitis, or a history of chronic or acute pancreatitis, as determined by the investigator
* Serum amylase >=3 ×ULN and/or serum lipase >=2 × ULN and/or subject is experiencing any symptoms possibly related to pancreatitis
* Prior use of a GLP-1R agonist or DPP-IV inhibitor within 6 months before Screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2013-02-23 (Actual); Primary Completion 2015-01-27 (Actual); Study Completion 2015-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- Japan (23):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Okuda I, Wilson TH, Yue L, Nakajima H, Carr MC, Tsuboi M, Nino A, Seino Y. Albiglutide, a weekly GLP-1 receptor agonist, improves glycemic parameters in Japanese patients with type 2 diabetes over 1 year when added to single oral antidiabetic drugs. Curr Med Res Opin. 2017 Mar;33(3):431-438. doi: 10.1080/03007995.2016.1261817. Epub 2016 Dec 21. PMID 27852119
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116170 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 360 participants with type 2 diabetes mellitus (T2DM) were planned and 374 participants were enrolled and analyzed in the Safety Population; the Safety Population and Intent-to-Treat Population were identical in this study.
Pre-assignment Details: Eligible participants entered a 2-week Screening Period; a 52-week Treatment Period and an 8-week Follow-up (FU) Period.
Groups:
- Albiglutide Plus (+) Background OAD (Sulfonylurea): Participants received current regimen of 30 milligrams (mg) albiglutide + sulfonylurea (with titration to 50 mg at Week 4 or later based on specific guidelines on glycemic control) through Week 52.
- Albiglutide Plus (+) Background OAD (Biguanide): Participants received current regimen of 30 mg albiglutide + biguanide (with titration to 50 mg at Week 4 or later based on specific guidelines on glycemic control) through Week 52.
- Albiglutide Plus (+) Background OAD (Glinide): Participants received current regimen of 30 mg albiglutide + glinide as a subcutaneous injection weekly (with titration to 50 mg at Week 4 or later based on specific guidelines on glycemic control) through Week 52.
- Albiglutide Plus (+) Background OAD (Thiazolidinedione): Participants received current regimen of 30 mg albiglutide + thiazolidinedione as a subcutaneous injection weekly (with titration to 50 mg at Week 4 or later based on specific guidelines on glycemic control) through Week 52.
- Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor): Participants received current regimen of 30 mg albiglutide + α-glucosidase inhibitor as a subcutaneous injection weekly (with titration to 50 mg at Week 4 or later based on specific guidelines on glycemic control) through Week 52.
Period: Overall Study
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Started | 120 | 67 | 65 | 61 | 61
Completing Treatment Period | 109 | 63 | 59 | 59 | 54
Completing Follow-up Period | 109 | 63 | 59 | 59 | 54
Completed | 109 | 63 | 59 | 59 | 54
Not Completed | 11 | 4 | 6 | 2 | 7
Not completed — Persistent Hyperglycemia | 0 | 0 | 1 | 0 | 0
Not completed — New Antidiabetic Medication | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 2 | 0 | 1 | 0 | 2
Not completed — Moved, transfer abroad, did not enter FU | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor) | Total
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 61 | 374
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (9.19) | 57.0 (8.55) | 55.7 (11.07) | 59.0 (10.54) | 57.4 (10.47) | 57.7 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 22 | 22 | 11 | 20 | 108
  Male | 87 | 45 | 43 | 50 | 41 | 266
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 120 | 67 | 65 | 61 | 61 | 374

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of non-serious AEs and SAEs. Non-serious hypoglycemia events are not included.
Time Frame: From Baseline through Week 52
Population: Safety Population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 61
Participants
  Any AE | 97 | 47 | 58 | 49 | 43
  Any SAE | 2 | 0 | 1 | 2 | 3

2. Primary Outcome: Number of Participants With Any Hypoglycemic Event
Description: Hypoglycemia events are defined with respect to low plasma glucose level, mostly accompanied by typical symptoms and/or assistance needed from third party with glucose administration. These events were reported by the investigators upon verification of the plasma glucose levels, symptoms and assistance recorded by the participants, and/or plasma glucose values obtained from laboratory evaluations.
Time Frame: From Baseline through Week 52
Population: Safety Population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 61
Participants | 17 | 1 | 4 | 2 | 0

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the value at Week 52 minus the value at Baseline. Participants who discontinued from study treatment before Week 52 had their last on-treatment, post-Baseline HbA1c observation carried forward for the analysis.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Last Observation Carried Forward) Population: all enrolled participants who received at least 1 dose of study medication and who had at least one HbA1c post-Baseline assessment.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 60
Percentage of HbA1c in the blood | -1.04 (0.657) | -0.94 (0.623) | -0.95 (0.836) | -1.42 (0.771) | -1.39 (0.770)

4. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Levels of HbA1c (i.e., the Percentage of Participants Achieving Treatment Goal of <6.5% and <7.0% at Week 52)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3 month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Participants who discontinued from study treatment before Week 52 had their last on-treatment, post-Baseline HbA1c observation carried forward for the analysis. Clinically meaningful levels of response in HbA1c are defined as <6.5% and <7.0%.
Time Frame: Week 52
Population: Intent-to-Treat (Last Observation Carried Forward) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 60
Percentage of participants
  HbA1c <6.5% | 20.0 | 26.9 | 24.6 | 45.9 | 26.2
  HbA1c <7.0% | 54.2 | 59.7 | 52.3 | 80.3 | 67.2

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: FPG is an indicator of efficacy. The Baseline FPG value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the FPG value at Week 52 minus the FPG value at Baseline. Participants who discontinued from study treatment before Week 52 had their last on-treatment, post-Baseline FPG observation carried forward for the analysis.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Last Observation Carried Forward) Population. Only those participants with valid post-Baseline results (within 14 days of last exposure to treatment) were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 59
Milligrams per deciliter (mg/dL) | -16.4 (28.52) | -24.3 (19.98) | -16.4 (30.37) | -32.1 (27.21) | -33.2 (28.38)

6. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline body weight value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the body weight value at Week 52 minus the value at Baseline. Participants who discontinued from study treatment before Week 52 had their last on-treatment, post-Baseline weight observation carried forward for the analysis.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Last Observation Carried Forward) Population
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 120 | 67 | 65 | 61 | 60
Kilograms (kg) | 0.25 (2.167) | -0.33 (2.082) | -0.04 (2.405) | 0.52 (2.823) | -0.13 (2.620)

7. Secondary Outcome: Time to Study Withdrawal Due to Hyperglycemia
Description: Participants who experienced persistent hyperglycemia after uptitration were to be withdrawn from the study. Hyperglycemia is defined as a fasting plasma glucose >=280 mg/dL (>=15.5 mmol/L) from >=Week 2 to <Week 12 or >=230 mg/dL (>=12.8 mmol/L) from >=Week 12 to <Week 52.
Time Frame: Week 52
Population: Intent-to-Treat (Last Observation Carried Forward) Population. Only participants who were withdrawn due to hyperglycemia were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Number analyzed (Participants) | 1 | 0 | 2 | 0 | 0
Weeks | 13.0 (NA) — There were too few events to provide an estimable standard deviation. |  | 16.5 (3.54) |  |

ADVERSE EVENTS:
Time Frame: On-therapy non-serious adverse events (AEs) and serious adverse events (SAEs) with an onset date on or after the start date of study treatment and within 56 days after the date of the last dose of study treatment, are summarized through Week 52.
Description: The non-serious AEs and SAEs are reported for the Safety Population, which comprised of all participants who received at least 1 dose of study treatment; par. underwent uptitration of albiglutide from 30 mg to 50 mg weekly based on glycemic parameters.
Arm/Group | Albiglutide Plus (+) Background OAD (Sulfonylurea) | Albiglutide Plus (+) Background OAD (Biguanide) | Albiglutide Plus (+) Background OAD (Glinide) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor)
Serious Adverse Events (participants affected / at risk) | 2/120 | 0/67 | 1/65 | 2/61 | 3/61
Other Adverse Events (participants affected / at risk) | 68/120 | 31/67 | 38/65 | 35/61 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Plus (+) Background OAD (Sulfonylurea) (N=120) | Albiglutide Plus (+) Background OAD (Biguanide) (N=67) | Albiglutide Plus (+) Background OAD (Glinide) (N=65) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) (N=61) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor) (N=61)
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Plus (+) Background OAD (Sulfonylurea) (N=120) | Albiglutide Plus (+) Background OAD (Biguanide) (N=67) | Albiglutide Plus (+) Background OAD (Glinide) (N=65) | Albiglutide Plus (+) Background OAD (Thiazolidinedione) (N=61) | Albiglutide Plus (+) Background OAD (α-Glucosidase Inhibitor) (N=61)
Nasopharyngitis (Infections and infestations) | 37 | 19 | 30 | 19 | 17
Constipation (Gastrointestinal disorders) | 15 | 1 | 4 | 5 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 1 | 4 | 2 | 0
Diabetic retinopathy (Eye disorders) | 8 | 3 | 0 | 5 | 4
Bronchitis (Infections and infestations) | 4 | 4 | 1 | 2 | 3
Pharyngitis (Infections and infestations) | 4 | 2 | 2 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 6 | 1 | 2 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 8 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.